CLINICAL TRIAL: NCT03314883
Title: Ultrasound Diaphragmatic Evaluation in Acute Hypoxic - Hypercapnic Respiratory Failure (ARF) Patients Undergoing Non Invasive Ventilation: A Pilot Feasibility Study
Brief Title: Diaphragmatic Ultrasound in Acute Hypoxic - Hypercapnic Respiratory Failure (ARF)
Acronym: DiaDea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Principal Investigator, MD of ICU staff, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 112/17
Record Dates: First submitted 2017-09-22; First posted 2017-10-19 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Acute Hypoxic - Hypercapnic Respiratory Failure (ARF)
Keywords: Ultrasound; Diaphragm; Non Invasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-US ARF (Experimental): Diaphragmatic evaluation, i.e thickening fraction (%) and excursion (millimeters), will be performed 3 times in the first two hours after acute hypoxic - hypercapnic respiratory failure (ARF) patients admission
  Interventions: Diagnostic Test: D-US ARF

INTERVENTIONS:
Diagnostic Test: D-US ARF — Diaphragm ultrasound evaluation in acute hypoxic - hypercapnic respiratory failure (ARF) patients undergoing non invasive ventilation, with regard to thickening (%) and excursion (millimeters)

SUMMARY:
Mortality of acute hypoxic - hypercapnic respiratory failure (ARF) patients underwent invasive mechanical ventilation is demonstrated to be higher than in patients who underwent only non invasive mechanical ventilation (NIV).

There is an increased need to detect more predictive factors for NIV failure, in order to better identify patients most at risk of facing negative outcomes.

The aim of this experimental pilot study is to evaluate the feasibility of the ultrasound of diaphragm in ARF patients underwent non invasive mechanical ventilation ( primary endpoint ).

Furthermore the secondary aim is to observe any relationship between diaphragmatic function (excursion), diaphragmatic thickening and the timing of arterial blood gases (ABGs) compensation in patients with ARF undergoing NIV treatment; additional outcomes are: correlation with dyspnea level, time of mechanical ventilation, NIV failure, rate of tracheostomy, length of stay in ICU and in-hospital and 90-day mortality.

DETAILED DESCRIPTION:
Inclusion criteria: respiratory failure resulting in respiratory acidosis to be treated with NIV, age> = 18 years

Exclusion criteria: acute pulmonary edema, coexisting interstitial pathologies, neuromuscular pathologies, thoracic cage's deformity, previous diaphragmatic paralysis, hemodynamic instability, intracranial hypertension, pregnancy, absolute contraindications to NIV, need for immediate intubation, recent thoracotomy, presence of pneumothorax or pneumomediastinum.

After patient's triage, transfer to Shock Room and primary assessment by emergency department staff ,diaphragmatic ultrasound is performed when NIV indication is given.

NIV is delivered with a facial mask; ventilation is set in NIV application, pressure support mode. Positive end expiratory pressure (PEEP) and Inspired oxygen fraction (FiO2) are adjusted to obtain a peripheral oxygen saturation (Spo2) between 88-92%. The pressure support is set to achieve a target volume of between 6-8 (ml / kg) and a respiratory rate < 30 respiratory acts per minute.

Respectively one and two hours after starting NIV, diaphragmatic ultrasonography and ABGs analysis are again performed.

NIV failure criteria are defined by the need for endotracheal intubation or by death.

Criteria for NIV failure: unchanging or worsening blood gases despite NIV; need to protect airways due to neurological deterioration or massive secretions; haemodynamic instability or major electrocardiographic abnormalities; uncontrolled dyspnea and NIV intolerance/ refusal.

General measures On admission clinical severity is recorded by Glasgow Coma Scale (GCS), Acute Physiology and Chronic Health Evaluation II Score (APACHE II).

ABGs values ( PH, arterial oxygen tension (paO2), arterial carbon dioxide tension (paCo2), paO2/FiO2, bicarbonates (HCO3), lactate) will be recorded before NIV, at 1 hour and 2 hours later.

Chest X-ray and peripheral blood sample (hemochrome with band cell count, C-reactive protein (CRP) and electrolytes) will be performed within 24 hours of admission.

The presence of pneumonia, sepsis and previous treatment with systemic or inhaled steroids will be recorded.

Diaphragm Ultrasound

Ultrasound evaluation of diaphragm function is performed on admission before starting NIV, 1 hour and 2 hours later.

Diaphragmatic function is assessed by a B-Mode ultrasound device connected to a linear probe ( 7-12 MHz) at the patient's bedside.

Measurements are performed on a patient in supine position with a recessed back angle between 20 and 40 degrees.

Probe position is set between 8th and 10th intercostal space on the mid axillary line to find the apposition zone of the diaphragm, where lung, diaphragm and abdominal parenchyma are identifiable.

Diaphragmatic thickness is measured at end-inspiration ( Ti) and end- expiration (Te).

The percentage change in diaphragmatic thickness (ΔTdi) is calculated as follows:

ΔTdi % = (Ti- Te) / Te * 100 Measurements are performed three times and the average value of the three measurements is considered.

Diaphragmatic excursion is also evaluated.

Statistical analysis As it is an experimental pilot feasibility study, 20 patients will be initially enrolled.

Descriptive statistics for continuous variables will be presented as median and interquartile. Non-parametric continuous variables will be evaluated by non-parametric Wilcoxon test (Mann-Whitney).

Categorical variables will be evaluated by chi-square or Fisher's test.

The influence of diaphragmatic thickening and muscle thickness on NIV failure, mortality and hospitalization's days wil be assessed through correlation analysis A P-value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure resulting in respiratory acidosis to be treated with NIV
* Age> = 18 years

Exclusion Criteria:

* acute pulmonary edema
* coexisting interstitial pathologies
* neuromuscular pathologies
* thoracic cage's deformity
* previous diaphragmatic paralysis
* hemodynamic instability
* intracranial hypertension
* pregnancy
* absolute contraindications to NIV
* need for immediate intubation,
* recent thoracotomy
* presence of pneumothorax or pneumomediastinum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of diaphragm ultrasound function evaluation (excursion and thickening) in acute hypoxic - hypercapnic respiratory failure (ARF) during the first two hours after emergency department admission. | 2 hours
  Ultrasound will be performed before starting NIV, after 1 and 2 two hours of NIV application

SECONDARY OUTCOMES:
Arterial blood carbon dioxide (PaCO2) compensation evaluation | 0 hour
  PaCO2 at time of starting NIV, after one hour from NIV application and after two hours of NIV application
Arterial blood carbon dioxide (PaCO2) compensation evaluation | 1 hour
  PaCO2 at time of starting NIV, after one hour from NIV application
Arterial blood carbon dioxide (PaCO2) compensation evaluation | 2 hours
  PaCO2 after two hours from NIV application
Monitoring diaphragmatic function in terms of thickening at 0 hour | 0 hour
  Diaphragmatic thickening (%) [(inspiratory thickness - expiratory thickness)]/expiratory thickness * 100
Monitoring diaphragmatic function in terms of thickening at 1 hour | 1 hour
  Diaphragmatic thickening (%) [(inspiratory thickness - expiratory thickness)]/expiratory thickness * 100
Monitoring diaphragmatic function in terms of thickening at 2 hours | 2 hours
  Diaphragmatic thickening (%) [(inspiratory thickness - expiratory thickness)]/expiratory thickness * 100
Monitoring diaphragmatic function in terms of excursion at 0 hour | 0 hour
  Diaphragmatic excursion (millimeters) computed as diaphragmatic displacement during breath
Monitoring diaphragmatic function in terms of excursion at 1 hour | 1 hour
  Diaphragmatic excursion (millimeters) computed as diaphragmatic displacement during breath
Monitoring diaphragmatic function in terms of excursion at 2 hours | 2 hours
  Diaphragmatic excursion (millimeters) computed as diaphragmatic displacement during breath
Days spent in intensive care unit | 28 days
  Amount of days spent in ICU
Days spent in in hospital | 90 days
  Amount of days spent in hospital
dyspnea level at 0 hour | 0 hour
  dyspnea level evaluated via visual analogical scale
dyspnea level at 1 hour | 1 hour
  dyspnea level evaluated via visual analogical scale
dyspnea level at 2 hours | 2 hours
  dyspnea level evaluated via visual analogical scale

OTHER OUTCOMES:
Relationship with mechanical ventilation length | 28 days
  mechanical ventilation length expressed in days for both invasive and non invasive ventilation
Mortality in intensive care unit | 28 days
  Number of death in intensive care unit
Tracheostomy | 28 days
  Rate of tracheostomy (ratio between number of tracheostomy in study group)
Relation with gravity index | 24 hours
  value of APACHE score in study population
Mortality in hospital | 90 days
  Number of death in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cammarota G, Sguazzotti I, Zanoni M, Messina A, Colombo D, Vignazia GL, Vetrugno L, Garofalo E, Bruni A, Navalesi P, Avanzi GC, Della Corte F, Volpicelli G, Vaschetto R. Diaphragmatic Ultrasound Assessment in Subjects With Acute Hypercapnic Respiratory Failure Admitted to the Emergency Department. Respir Care. 2019 Dec;64(12):1469-1477. doi: 10.4187/respcare.06803. Epub 2019 Aug 27. PMID 31455684